CLINICAL TRIAL: NCT03652259
Title: A Single-Center, Open-Label, Systemic Gene Delivery Study to Evaluate the Safety, Tolerability, and Efficacy of SRP-9003 Administered by Systemic Infusion in Subjects With LGMD2E (β-Sarcoglycan Deficiency)
Brief Title: Gene Delivery Clinical Trial of SRP-9003 (Bidridistrogene Xeboparvovec) for Participants With Limb-Girdle Muscular Dystrophy, Type 2E (LGMD2E) (Beta-Sarcoglycan Deficiency)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is being terminated due to a business decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9003-101; IRB17-00253 (Other: Sarepta Therapeutics)
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Limb-Girdle Muscular Dystrophy, Type 2E
Keywords: limb girdle muscular dystrophy; LGMD2E; beta-sarcoglycan; gene transfer; adeno-associated virus; LGMDR4
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2E; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: SRP-9003 (Experimental): Participants will receive a single intravenous (IV) infusion of SRP-9003 at a prespecified dose.
  Interventions: Genetic: SRP-9003
- Cohort 2: SRP-9003 (Experimental): Participants will receive a single IV infusion of SRP-9003. Dose will be determined based on the findings from Cohort 1.
  Interventions: Genetic: SRP-9003

INTERVENTIONS:
Genetic: SRP-9003 — SRP-9003 will be administered through a single systemic injection.
  Other Names: LGMD2E vector; bidridistrogene xeboparvovec

SUMMARY:
The proposed clinical trial is the first-in-human, single-center, open-label, gene delivery study of SRP-9003 (bidridistrogene xeboparvovec) in participants with LGMD2E.

ELIGIBILITY:
INCLUSION CRITERIA

* Males or females of any ethnic group
* β-SG deoxyribonucleic acid (DNA) gene mutations at both alleles
* Weakness demonstrated based on history of difficulty in running, jumping and climbing stairs
* A 100 meter walk/run (MWR) test result: ≥40 % of predicted for age-, height-, gender-, and weight-matched healthy controls at the screening visit

EXCLUSION CRITERIA

* Active viral infection based on clinical observations
* Cardiac magnetic resonance imaging (MRI) determined left ventricular ejection fraction (LVEF) <40%
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Abnormal laboratory values considered clinically significant
* Concomitant illness or requirement for chronic drug treatment that, in the opinion of the Principal Investigator, creates unnecessary risks for gene transfer.

Other inclusion/exclusion criteria apply.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs) | Baseline up to 7 years

SECONDARY OUTCOMES:
Change From Baseline in Quantity of Beta-Sarcoglycan (β-SG) Protein Expression at Day 60, as Measured by Western Blot | Baseline, Day 60
  β-SG gene expression levels will be quantified by Western Blot and compared between pre and post muscle biopsies.
Change From Baseline in Quantity of β-SG Protein Expression at Day 60, as Measured by Immunofluorescence | Baseline, Day 60
  β-SG gene expression levels will be quantified by immunofluorescence and compared between pre and post muscle biopsies.
Change From Baseline in Quantity of β-SG Protein Expression at Day 60, as Measured by Immunohistochemistry Percent B-SG Positive Fibers | Baseline, Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Mendell JR, Pozsgai ER, Lewis S, Griffin DA, Lowes LP, Alfano LN, Lehman KJ, Church K, Reash NF, Iammarino MA, Sabo B, Potter R, Neuhaus S, Li X, Stevenson H, Rodino-Klapac LR. Gene therapy with bidridistrogene xeboparvovec for limb-girdle muscular dystrophy type 2E/R4: phase 1/2 trial results. Nat Med. 2024 Jan;30(1):199-206. doi: 10.1038/s41591-023-02730-9. Epub 2024 Jan 4. PMID 38177855